CLINICAL TRIAL: NCT05370027
Title: Investigation of the Effect of Unilateral Right, Unilateral Left and Bilateral Applications of Transcutaneous Auricular Vagus Nerve Stimulation on Autonomic Nervous System Activity in Healthy People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Berkay Eren PEHLIVANOGLU, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BahcesehirU_B.Pehlivanoglu001
Record Dates: First submitted 2022-04-26; First posted 2022-05-11 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Health, Subjective
Keywords: vagus nerve; vagus nerve stimulation; transcutaneous auricular vagus nerve stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1st Group (Experimental): With the vagustim device, the application will be made first from the left ear. Then, a 48-hour break will be taken and the application will be made from the right ear. Then, the application will be performed on both ears with a 48-hour break.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- 2nd Group (Experimental): With the vagustim device, the application will be made first from the left ear. Then, a 48-hour break will be made and the application will be made from both ears. Then, the application will be performed on the right ear with a break for 48 hours.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- 3rd Group (Experimental): With the vagustim device, the application will be made first from the right ear. Then, a 48-hour break will be taken and the application will be made from the left ear. Then, the application will be performed on both ears with a 48-hour break.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- 4th Group (Experimental): With the vagustim device, the application will be made first from the right ear. Then, a 48-hour break will be made and the application will be made from both ears. Then, the application will be performed on the left ear with a break for 48 hours.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- 5th Group (Experimental): With the vagustim device, the application will be made from both ears first. Then, a 48-hour break will be made and the application will be made from the left ear. Then, the application will be performed on the right ear with a break for 48 hours.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- 6th Group (Experimental): With the vagustim device, the application will be made from both ears first. Then, a 48-hour break will be made and the application will be made from the right ear. Then, the application will be performed on the left ear with a break for 48 hours.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Vagus nerve stimulation will be applied with the Vagustim device for 20 (10+10) minutes, with a biphasic frequency, a frequency of 10 Hz, a pulse width of 300 μs in Modulation mode, and a constant current intensity where the participant feels the current comfortably.

SUMMARY:
The vagus nerve is one of the main components of the parasympathetic nervous system, which oversees a wide variety of important bodily functions, including mood control, immune response, digestion, and heart rate. It is the tenth cranial nerve originating from the medulla oblongata in the central nervous system and is the longest cranial nerve. It starts from the medulla and progresses to the colon. It mainly innervates the thoracic and abdominal organs. It has an obvious effect on the autonomic nervous system, especially on parasympathetic activity. When the literature is examined, it has been proven by various studies that vagus nerve stimulation has effects on the regulation of the autonomic system. Vagus nerve stimulation with different methods has been investigated over the years and the effectiveness of several different methods has been proven. There are both invasive and non-invasive (transcutaneous) techniques for vagus nerve stimulation. The first experiments were developed on invasive applications, and then non-invasive applications began to emerge.

Today, the most used devices and stimulation models were approved by the FDA in the 1990s for use in patients with drug-resistant epilepsy. In the middle of the first decade of the 2000s, the FDA approved the use of these devices for drug-resistant depression. These application methods have therapeutic effects for a wide variety of conditions, including heart failure, obesity, migraine, Alzheimer's, inflammation, chronic pain, and tinnitus. Invasive intervention is not necessary to perform this procedure. Direct stimulation of afferent nerve fibers in the ear can produce a similar effect without surgical intervention. Non-invasive vagus nerve stimulation may affect human physiology and be a simple and inexpensive alternative to invasive vagus stimulation. It has been shown on different subjects that non-invasive stimulation of the tragus in the ear increases the activation in the parasympathetic system and decreases the sympathetic activity. This indicates that tragus stimulation may be a viable treatment for some disorders in which autonomic activity is compromised.

While the general mechanism has been explained in this way, there is no definite information in the literature about which ear from the right single ear, double ear or left single ear will be applied in Transcutaneous Auricular Vagus Nerve Stimulation applications. While specifying the application techniques, an objective scientific study about whether there is a difference between Unilateral Right, Unilateral Left and Bilateral Applications or which of them gives more effective results will be a guide for further studies. The purpose of the study, planning to carry out is to seek an answer to one of the questions that come to mind for standardization. The main question we seek to answer is whether there is a difference between Unilateral Right, Unilateral Left and Bilateral Applications while specifying the application techniques, or which of them gives more effective results. This studies main goal is to set up this study in order to seek answers about which application style will produce results and to provide a guide for further studies.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Have signed the informed consent form
* The volunteer has no disease before or during the study
* Absence of menstrual cycle period in female volunteers
* The subject did not drink alcohol 24 hours before the study

Exclusion Criteria:

* Cases unwilling to continue the study.
* Having a respiratory disease and starting to use drugs
* Having a disease related to the cardiac system and starting to use drugs
* The presence of any chronic disease and the use of a drug related to it

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | Up to 1 week
  Omron Hem 7321 E M6 device will be used to measure heart rate
Systolic and Diastolic Blood Pressure | Up to 1 week
  Omron Hem 7321 E M6 device will be used to measure Systolic and Diastolic Blood Pressure
Evaluation of Galvanic Skin Resistance | Up to 1 week
  Bogazici University GSR device will be used to measure Galvanic Skin Resistance
Heart Rate Variability | Up to 1 week
  Elite HRV device will be used to measure Heart Rate Variability

IPD SHARING:
Plan to Share IPD: Undecided